CLINICAL TRIAL: NCT04132440
Title: Patient and Physician Perspectives on Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Patient and Physician Perspectives on Non-Alcoholic Fatty Liver Disease
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-0262; NCI-2019-05886 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0262 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-10-04; First posted 2019-10-18 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Nonalcoholic Fatty Liver Disease; Physician
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, interview): Patients and physicians complete a questionnaire over 5 minutes and an interview over 30-45 minutes about thoughts on NAFLD, including what they know about NAFLD and its diagnosis, management, and monitoring, and other thoughts on NAFLD.
  Interventions: Other: Interview; Other: Questionnaire Administration

INTERVENTIONS:
Other: Interview — Complete interview
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This trial studies patient and physician perspectives on non-alcoholic fatty liver disease. Using questionnaires and interviews, this trial may help researchers understand physicians' knowledge about the diagnosis, prognosis, treatment and management of non-alcoholic fatty liver disease, as well as gain an in-depth understanding of Hispanic patients' perceptions about the disease and investigate how cultural factors may play a role in its diagnosis, treatment and management.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Explore the perceptions of non-alcoholic fatty liver disease (NAFLD), including knowledge, current practices for diagnosis and management, and additional disease-related perceptions amongst both primary care physicians.

II. Explore the perceptions of NAFLD, including knowledge, diagnosis and management, and additional disease-related perceptions amongst Hispanic patients.

OUTLINE:

Patients and physicians complete a questionnaire over 5 minutes and an interview over 30-45 minutes about thoughts on NAFLD, including what they know about NAFLD and its diagnosis, management, and monitoring, and other thoughts on NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Be a self-reported practicing physician, who is a primary care physician (internal medicine, family medicine, etc.)
* Self-reported Hispanic ethnicity from the Greater Houston Metropolitan Area (patient)
* Have been diagnosed with NAFLD by a doctor (patient)
* Be an adult >/= 18 (patient)
* Able to speak English (patient)

Exclusion Criteria

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hispanic patients with NAFLD from the Greater Houston Metropolitan Area and practicing physicians, who are primary care physicians (internal medicine, family medicine, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Explore the perceptions of NAFLD, including knowledge, current practices for diagnosis and management, and additional disease-related perceptions amongst both primary care physicians (Questionnaire) | Up to 1 year
Explore the perceptions of NAFLD, including knowledge, diagnosis and management, and additional disease-related perceptions amongst Hispanic patients. (Questionnaire) | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lorna McNeill, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org